CLINICAL TRIAL: NCT04245644
Title: Efficacy of Chemopreventive Agents on Disease-free and Overall Survival in Patients With Pancreatic Ductal Adenocarcinoma: The CAOS Study
Acronym: CAOS
Status: Active, not recruiting | Type: Observational
Sponsor: Massimo Falconi (Other)
Responsible Party: Sponsor-Investigator, Massimo Falconi, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: CAOS
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Disease Free Survival; Overall Survival; Pancreatic Cancer
Keywords: aspirin,; metformin; statin; ACE-inhibitors; beta-blockers; pancreatic cancer; survival
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Aspirin; Metformin; Angiotensin-Converting Enzyme Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: use of targeted drugs such as aspirin, B-Blockers, Metformin, ACE-inhibitors, Statins — enrolled patients will be asked details regarding their daily drug use, before and after diagnosis of pancreatic cancer

SUMMARY:
The evidence on the value of aspirin, statins, metformin, beta-blocking ACE inhibitors agents as chemopreventive agents in patients with pancreatic ductal adenocarcinoma is limited.

The aim of this study is to assess whether regular use of aspirin, statins, metformin, angiotensin converting enzyme (ACE)-inhibitors and beta-blocking agents use, before diagnosis, after surgery and in neo-adjuvant treatment setting, can increase rate of disease-free survival (DFS) and overall survival (OS) in participants with pancreatic ductal adenocarcinoma. The secondary aim is to evaluate if there is any difference in terms of "chemoprevention" between aspirin, statins, metformin and beta-blocking as chemopreventive agents, and if their prolonged daily use can positively influence the chemopreventive action.

400 patients with the following inclusion criteria will be enrolled in 3 years:

1. cytological or histological diagnosis of pancreatic ductal adenocarcinoma in any portion of the gland, with or without metastases in other sites
2. patient age between 18 and 90 years
3. any medicine or drug in the daily patient therapy
4. Patients undergone to primary chemoradiotherapy or surgical resection, followed by adjuvant therapy or preceded by neoadjuvant chemoradiotherapy, are included in the study Anamnestic, clinical and pathological data, included data on the aspirin, statins, metformin, angiotensin converting enzyme (ACE)-inhibitors and beta-blocking agents assumption will be collected during the first visit with the surgeon. A database managed by a dedicated data manager will be created to collect and analyse data.

Patients will be followed for at least 24 months The study will last overall 5 years.

DETAILED DESCRIPTION:
Sample size and Population

This study is designed as a monocentric observational prospective study. In a recent study [9] authors found that the use of low-dose aspirin before and after a diagnosis of pancreatic cancer reduces of 32% the risk of recurrence (Hazard ratio HR=0.68, p<0.01). On the basis of this study and considering that the effect of other drugs as chemopreventive agentsw will be studies, the estimate required sample size to achieve 90% power to detect at least 28% reduction in a hazard of the "drug users" group, by using a two-sided 0.05-level log-rank test, is 400. Therefore, from February 2019 to February 2022, 400 patients with a diagnosis of pancreatic ductal adenocarcinoma at any stage meeting the following inclusion criteria are expected to be enrolled. Median follow-up is estimated to be 24 months after the first disease diagnosis.

Data collection methods

Anamnestic, clinical and pathological data, included data on the aspirin, statins, metformin, angiotensin converting enzyme (ACE)-inhibitors and beta-blocking agents assumption will be collected during the first visit with the surgeon. A database managed by a dedicated data manager will be created to collect and analyse data. The PI will be responsible of the data security.

Statistical analysis

Association between variables will be assessed using the Chi Squared test (or Fisher's exact text where appropriate) for categorical variables and the Spearman's correlation for scale variables. DFS and OS will be estimated using Kaplan-Mayer method and Log Rank tests will be used to evaluate the difference between survival curves. The impact of aspirin, statins, metformin, angiotensin converting enzyme (ACE)-inhibitors and beta-blocking agents on the risk of recurrence will be estimated using Cox regression models. Variables resulting significant (p value <0.05) at univariate analysis or variables which are known prognostic/risk factors will be included in the multivariable regression models. A p value of <0.05 will be considered statistically significant. Statistical analysis will be conducted using SPSS v23 (IBM, Armonk, New York, USA) and R v3.3.0 (https://cran.r-project.org).

ELIGIBILITY:
Inclusion Criteria:

1. cytological or histological diagnosis of pancreatic ductal adenocarcinoma in any portion of the glande, with or without metastases in other sites
2. patient age between 18 and 90 years
3. any medicine or drug in the daily patient therapy
4. Patients undergone to primary chemoradiotherapy or surgical resection, followed by adjuvant therapy or preceded by neoadjuvant chemoradiotherapy, are included in the study

Exclusion Criteria:

1. age under 18 years
2. lack of cytological or histological diagnosis of pancreatic ductal adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with a diagnosis of pancreatic ductal adenocarcinoma in any portion of the glande, with or without metastases in other sites
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | two-years follow-up
  probability of recurrence or progression of disease in patients on regular treatment with targeted drugs compared with non-users
Overall survival | two-years follow-up
  risk of death for disease in patients on regular treatment with targeted drugs compared with non-users

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No